CLINICAL TRIAL: NCT01212198
Title: Clinical Research Center For Type 2 Diabetes Mellitus - Observational Cohort Study of Type 2 Diabetes Mellitus
Brief Title: Korea National Diabetes Program
Acronym: KNDP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Korea University Guro Hospital (Other); Hanyang University (Other); Inha University Hospital (Other); Ajou University (Other); East West Neo Medical Center (Other); Pusan National University Hospital (Other); Gachon University Gil Medical Center (Other); Cheil General Hospital and Women's Healthcare Center (Other); Yeungnam University Hospital (Other); Inje University (Other); Kangdong Sacred Heart Hospital (Other); Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Young-Seol Kim, MD, PhD, Kyunghee University Medical Center
Other Study IDs: KNDP-KMC-0505
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-09

CONDITIONS: Type 2 Diabetes Mellitus; Diagnosis; Treatment; Prevention; Complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Korean type 2 diabetic patients
- Koreans at high risk for diabetes
- Korean gestational diabetic patients

SUMMARY:
This is an observational study done by creating a cohort of Korean patients with diabetes and those at high risk of developing diabetes. By the creation of this cohort we aim to establish efficient preventive, diagnostic, and therapeutic measures based on the characteristics of Korean patients with diabetes, and by doing so, we hope to ultimately decrease our country's diabetes-related-mortality and increase the quality of life of patients with type 2 diabetes.

DETAILED DESCRIPTION:
It is estimated that in 20 years the number of patients with diabetes will be over 6 million. Therefore the importance of diagnosis, treatment, and prevention of diabetes needs no further emphasis. At the moment, current studies demonstrate that mortality has increased twofold in the last 10 years due to lack of adequate control, and that medical expenses related to diabetes is increasing. Therefore, the necessity to find means for effective prevention and management of diabetes seems pressing.

However, unfortunately, in Korea, results of systematic clinical trials carried out in the Korean population are not available. All the currently available management guidelines have been formulated based on the results of clinical trials carried out in other populations, on patients with perhaps different characteristics compared to ours. There are quite a number of problems in applying these guidelines to our patients.

This study's purpose is to create a basis on which we could establish effective prevention, diagnosis, and therapeutic plan based on specific characteristics of Korean patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

(Group 1:Diagnostic criteria for type 2 diabetes based on ADA 2004 guidelines)

* random plasma glucose >200mg/dL + symptoms such as polyuria, polydipsia, unexplained weight loss
* fasting plasma glucose >126 mg/dL or 75g oral glucose tolerance test (OGTT) 2h plasma glucose >200 mg/dL (Group 2: High risk for diabetes based on ADA 2004 guidelines)
* IFG: fasting plasma glucose 100-125 mg/dL and 75g OGTT 2h plasma glucose <140 mg/dL
* IGT: fasting plasma glucose <100 mg/dL and 75g OGTT 2h plasma glucose 140-199 mg/dL (Group 3: Gestational Diabetes based on ADA 2004 guidelines)
* 50g OGTT 1h plasma glucose >140 mg/dl
* 100g OGTT fasting plasma glucose >95 mg/dl, 1h plasma glucose >180 mg/dl, 2h plasma glucose >155 mg/dL, 3h plasma glucose >140 mg/dL

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients with type 2 diabetes, Koreans at high risk for diabetes, Korean patients with gestational diabetes
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2005-05; Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Specific characteristics of Korean type 2 diabetic patients | up to 10 years
  The investigators will investigate the characteristics of Korean type 2 diabetic patient.
  First planning time frame is up to 10 years, but this time frame can be needed, if needed. (If we need the extension of study duration, new informed consent will be gotten from patients)
Diabetes complications incidence and mortality in Korean type 2 diabetic patients | up to 10 years
  The investigators will investigate the characteristics of Korean type 2 diabetic patient.
  First planning time frame is up to 10 years, but this time frame can be needed, if needed. (If we need the extension of study duration, new informed consent will be gotten from patients)
Investigation of Korean type 2 diabetic patients' lifestyle | up to 10 years
  The investigators will investigate the characteristics of Korean type 2 diabetic patient.
  First planning time frame is up to 10 years, but this time frame can be needed, if needed. (If we need the extension of study duration, new informed consent will be gotten from patients)
Economic evaluation of Korean type 2 diabetic patients | up to 10 years
  The investigators will investigate the characteristics of Korean type 2 diabetic patient.
  First planning time frame is up to 10 years, but this time frame can be needed, if needed. (If we need the extension of study duration, new informed consent will be gotten from patients)
Incidence of diabetes in patients with high risk for diabetes and gestational diabetes in Koreans | up to 10 years
  The investigators will investigate the characteristics of Korean type 2 diabetic patient.
  First planning time frame is up to 10 years, but this time frame can be needed, if needed. (If we need the extension of study duration, new informed consent will be gotten from patients)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Seol Kim, MD, PhD, Principal Investigator — Kyunghee University Medical Center
Locations (12):
- South Korea (12):
  - Hanyang University Medical Center, Guri-si, Kyunggi
  - Gachon University Gil Hospital, Incheon, Namdong
  - Yeungnam University Medical Center, Daegu
  - Inha University Hospital, Incheon
  - Pusan National University Hospital, Pusan
  - Cheil General Hospital, Seoul
  - Kyunghee University Medical Center, Seoul
  - Kangdong Sacred Heart Hospital Hallym University, Seoul
  - Inje University Sanggye-Paik Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University East West Neo Medical Center, Seoul
  - Ajou University Medical Center, Suwon

REFERENCES:
- [Derived] Kim SH, Hong SB, Suh YJ, Choi YJ, Nam M, Lee HW, Park IeB, Chon S, Woo JT, Baik SH, Park Y, Kim DJ, Lee KW, Kim YS; KNDP Study Group. Association between nutrient intake and obesity in type 2 diabetic patients from the Korean National Diabetes Program: a cross-sectional study. J Korean Med Sci. 2012 Oct;27(10):1188-95. doi: 10.3346/jkms.2012.27.10.1188. Epub 2012 Oct 2. PMID 23091316
- [Derived] Choi KM, Hwang SY, Hong HC, Yang SJ, Choi HY, Yoo HJ, Lee KW, Nam MS, Park YS, Woo JT, Kim YS, Choi DS, Youn BS, Baik SH. C1q/TNF-related protein-3 (CTRP-3) and pigment epithelium-derived factor (PEDF) concentrations in patients with type 2 diabetes and metabolic syndrome. Diabetes. 2012 Nov;61(11):2932-6. doi: 10.2337/db12-0217. Epub 2012 Jul 26. PMID 22837306